CLINICAL TRIAL: NCT00749437
Title: Feasibility of 3-D Conformal Accelerated Partial Breast Irradiation (APBI) for Early Stage, Node Negative Breast Cancer Patients Using Acculoc Fiducial Markers: A Phase I Trial
Brief Title: Radiation Therapy Using Gold Markers in Treating Women With Early-Stage Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 040801; P30CA072720 (NIH); CINJ-040801; CINJ-0220080173
Record Dates: First submitted 2008-09-06; First posted 2008-09-09 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; ductal breast carcinoma in situ; invasive ductal breast carcinoma; medullary ductal breast carcinoma with lymphocytic infiltrate; papillary ductal breast carcinoma; tubular ductal breast carcinoma; mucinous ductal breast carcinoma; breast cancer in situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Carcinoma, Ductal, Breast; Breast Carcinoma In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: 3-dimensional conformal accelerated partial breast irradiation — Accelerated partial breast irradiation following lumpectomy with placement of Acculoc fiducial markers.

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Placing gold markers in the area where the tumor was removed may help doctors better direct radiation therapy and help reduce the risk of cancer recurrence.

PURPOSE: This phase I trial is studying how well radiation therapy using gold markers works in treating women with early-stage breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if the delivery of external-beam accelerated partial breast irradiation (APBI) based on gold fiducial markers is more accurate when compared to the delivery of radiotherapy based on bony anatomy in women with early-stage, node-negative breast cancer.

Secondary

* To assess the migration of fiducial markers during a course of APBI.
* To quantify the change in the volume of the seroma (lumpectomy) cavity during a course of APBI.
* To compare overall operative time for suturing fiducial markers into place vs current standard method of placing surgical clips.

OUTLINE: Patients undergo planned lumpectomy with gold fiducial marker placement (if procedure not already performed). Patients who meet the post lumpectomy criteria for continue treatment in this study proceed to accelerated partial breast irradiation (APBI). Between 15-80 days after surgery, patients undergo 3-dimensional APBI (may be intensity-modulated radiotherapy) using CT-guided planning (with gold fiducial markers placed at lumpectomy) once daily, 5 days a week, for 15 days.

Patients undergo fluoroscopy weekly to determine real-time movement of bony anatomy and fiducial markers and cone-beam CT weekly to determine any change in volume of seroma cavity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Histologically confirmed ductal carcinoma in situ or invasive carcinoma of the breast (including ductal, medullary, papillary, colloid [mucinous], or tubular histologies) meeting all of the following criteria:

  * AJCC stage 0, I, or II (Tis, T1N0, or T2N0) disease with a lesion ≤ 3 cm treated with lumpectomy and either sentinel node biopsy or axillary dissection (if invasive carcinoma is present)
  * Unifocal breast cancer (i.e., single focus that can be encompassed by one lumpectomy)
* Underwent or plan to undergo lumpectomy with placement of gold fiducial markers (markers placed concurrently with the surgery or on a later date)

  * Patients who has underwent lumpectomy must meet all of the following criteria:

    * Must be enrolled between 14-60 days from date of last surgery, and radiation must start within 15-80 days of date of last surgery
    * Four to six gold fiducial markers placed in the tumor bed, delineating the margins of the lumpectomy cavity
    * Negative, inked histologic margins of lumpectomy (> 1 mm) or re-excision specimen to be confirmed prior to radiation

      * Margins are unacceptable if there is invasive or non-invasive tumor within 1 mm of the inked margin
* Negative post-excision mammography if malignancy-associated microcalcifications were initially present
* Hormone receptor status not specified

Exclusion criteria:

* Evidence of suspicious microcalcifications in the breast prior to the start of radiation
* One or more positive axillary nodes or positive sentinel biopsy
* Distant metastases
* Invasive or extensive in-situ lobular carcinoma or non-epithelial breast malignancies such as sarcoma or lymphoma
* Proven multicentric carcinoma (tumors in different quadrants of the breast or tumor separated by at least 4 cm) with other clinically or radiographically suspicious areas in the ipsilateral breast unless confirmed to be negative for malignancy by biopsy
* Palpable or radiographically suspicious contralateral axillary, supraclavicular, infraclavicular, or internal mammary nodes, unless there is histologic confirmation that these nodes are negative for tumor
* Paget's disease of the nipple
* Skin involvement, regardless of tumor size

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* ECOG performance status 0-1
* Life expectancy ≥ 2 years
* Not pregnant or nursing
* No prior treated breast carcinoma within the past 5 years
* No collagen vascular diseases, specifically systemic lupus erythematosus, scleroderma, or dermatomyositis
* No co-existing medical conditions
* No patients with medical conditions that would preclude compliance with the trial, as determined by the investigator
* No other malignancy, except non-melanomatous skin cancer, within the past 5 years

  * Disease-free interval from any prior carcinoma must be continuous
* No breast technically unsuitable for radiotherapy

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Concurrent tamoxifen citrate, anastrozole, or other hormonal therapy allowed
* Future chemotherapy allowed provided it is administered after the APBI and begins no earlier than 2 weeks after completion of radiotherapy
* No tylectomies so extensive that the cosmetic result is low or poor prior to radiation
* No prior radiation to the ipsilateral breast
* No prior non-hormonal therapy or radiotherapy for this disease
* No chemotherapy in the past 2 weeks
* No concurrent chemotherapy, immunotherapy, or experimental medications

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-10; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Amount of the shifts of the radiation fields based on bony anatomy as compared to that of gold fiducial markers | During radiation therapy

SECONDARY OUTCOMES:
Movement of the fiducial markers themselves and the change in volume of the seroma cavity during a 15-fraction course of accelerated radiotherapy compared with the pre-radiation volume | During radiation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Bruce G. Haffty, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States